CLINICAL TRIAL: NCT02006290
Title: A Phase 1b, Randomized, Subject And Investigator-Blinded, Sponsor-Open, Placebo Controlled, Cross-Over Efficacy, Safety And Tolerability Study Of Single Oral Split Dose Administration Of PF-06412562 In Subjects With Parkinson's Disease
Brief Title: Efficacy, Safety And Tolerability Study In Subjects With Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B7441003
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: PF-06412562
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-06412562 — single oral split dose 30+20 mg QD
  Arms: 1
Drug: Placebo — tablet, matching placebo, QD
  Arms: 2

SUMMARY:
The B7441003 study will assess PF-06412562 for motor benefit in Parkinson's disease subjects. Safety, tolerability and PK of PF-06412562 in Parkinson's disease subjects will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with a diagnosis of idiopathic Parkinson's disease.
* Daily L-dopa dose between 300 and 1200 mg.
* MBRS score >1.

Exclusion Criteria:

* Surgical intervention for Parkinson's disease.
* History of troublesome dyskinesias.
* Any significant AXIS I psychiatric disease.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Finger tapping speed | 12 hours
  maximum percent improvement from baseline in finger tapping speed as measured by the Kinesia Technology

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 0, 0.5, 1, 2, 4, 5,8,12, 24 hours
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0, 0.5, 1, 2, 4, 0, 0.5, 1, 2, 4, 8, 12, 24 hours
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0, 0.5, 1, 2, 4, 0, 0.5, 1, 2, 4, 8, 12, 24 hours
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Apparent Oral Clearance (CL/F) | 0, 0.5, 1, 2, 4, 0, 0.5, 1, 2, 4, 8, 12, 24 hours
Apparent Volume of Distribution (Vz/F) | 0, 0.5, 1, 2, 4, 8, 12, 24 hours
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Plasma Decay Half-Life (t1/2) | 0, 0.5, 1, 2, 4, 8, 12, 24 hours
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Mean Residence Time (MRT) | 0, 0.5, 1, 2, 4, 8, 12, 24 hours
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Number of Participants with categorical scores on the Columbia Suicide Severity Rating Scale (C-SSRS) | 24 hours
  C-SSRS assessed whether participant experienced following: completed suicide (1), suicide attempt (2) (response of "Yes" on "actual attempt"), preparatory acts toward imminent suicidal behavior (3)("Yes" on "preparatory acts or behavior"), suicidal ideation (4) ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent), any suicidal behavior or ideation, self-injurious behavior (7)("Yes" on "Has subject engaged in non-suicidal self-injurious behavior").

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - Pfizer Investigational Site, Aventura, Florida
  - Pfizer Investigational Site, Baco Raton, Florida
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, Bingham Farms, Michigan
  - Pfizer Investigational Site, Raleigh, North Carolina

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7441003